CLINICAL TRIAL: NCT06930222
Title: The Investigation of Predicting Mortality and Morbidity in Patients Admitted to Intensive Care Unit With Thoracic Trauma Using Selected Biomarkers and Parameters
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Suleyman Sencer CELİK, RESEARCH ASSISTANT, Suleyman Demirel University
Other Study IDs: SENCER-CELIK-001
Record Dates: First submitted 2025-01-03; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Thorax Traumas
Keywords: thorax trauma; ROX index; Surfactant-d
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — Hemogram Biochemical markers arterial blood gas analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- thorax trauma patients: thorax trauma patients admitted to icu
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — blood samples obtained for 3 different days, limited to 5cc

SUMMARY:
This prospective study aimed to predict morbidity and mortality after thoracic trauma in intensive care unit evaluated clinical and biochemical data of 50 intensive care unit patients. The research examined demographic factors such as gender, age, and smoking status, trauma scoring systems like ISS and RTS as well as biomarkers such as Surfactant-d and oxygenation parameters including the ROX index, PaO₂/FiO₂ ratio and FiO₂.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thoracic trauma between the ages of 18-85
* Patients who have been monitored in intensive care for at least 1 week

Exclusion Criteria:

* Being outside the age range of 18-85
* Pregnant patients
* Patients whose intensive care follow-up lasted less than 1 week
* Patients who do not want to be included in the study
* Patients with a lung malignancy diagnosis before admission

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thoracic trauma admitted to icu
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Mortality Prediction Using ROX Index in Thoracic Trauma Patients | Measurements taken on day 1, day 3, and day 7 of hospitalization, following ICU admission.
  To evaluate the predictive ability of the ROX index (unit: cmH₂O/L/s) for mortality in thoracic trauma patients. ROX index values were recorded at 1st, 3rd, and 7th days of hospitalization using standard clinical monitoring and ventilatory support parameters. Trends were analyzed in relation to survival outcomes.
Mortality Prediction Using SP-D Levels in Thoracic Trauma Patients | Measurements taken on day 1, day 3, and day 7 of hospitalization, following ICU admission.
  To assess the prognostic value of Surfactant Protein D (SP-D) levels (unit: ng/mL) for mortality prediction in thoracic trauma patients. SP-D levels were measured using an ELISA assay (Elabscience® Human Pulmonary Surfactant-associated Protein-D ELISA Kit) at 1st, 3rd, and 7th days to evaluate trends and correlations with survival outcomes.

SECONDARY OUTCOMES:
Predictive Value of APACHE II Score in Mortality | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  To analyze the effectiveness of the APACHE II score (range: 0-71; higher scores indicate worse outcomes) in predicting mortality in thoracic trauma patients. APACHE II scores were calculated based on clinical and laboratory parameters, including vital signs, blood gas values, and organ dysfunction markers at 1st, 3rd, and 7th days.
Predictive Value of SOFA Score in Mortality | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  To evaluate the prognostic accuracy of the Sequential Organ Failure Assessment (SOFA) score (range: 0-24; higher scores indicate worse outcomes) in thoracic trauma patients. SOFA scores were determined based on respiratory, cardiovascular, hepatic, coagulation, renal, and neurological functions at 1st, 3rd, and 7th days.
Predictive Value of TRISS Score in Mortality | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  To examine the relationship between Trauma and Injury Severity Score (TRISS) (range: 0-100%; higher scores indicate better survival probability) and survival outcomes in thoracic trauma patients. TRISS scores were calculated using physiological and anatomical injury severity data at 1st, 3rd, and 7th days.
Predictive Value of RTS Score in Mortality | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  To assess the relationship between Revised Trauma Score (RTS) (range: 0-7.84; higher scores indicate better prognosis) and mortality risk in thoracic trauma patients. RTS scores were calculated using Glasgow Coma Scale, systolic blood pressure, and respiratory rate values at 1st, 3rd, and 7th days.
CRP Levels and Mortality Prediction | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  To evaluate the association between C-reactive protein (CRP) levels (unit: mg/L) and mortality in thoracic trauma patients.
Procalcitonin Levels and Mortality Prediction | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  To analyze the prognostic value of procalcitonin (unit: ng/mL) levels in mortality prediction among thoracic trauma patients.

OTHER OUTCOMES:
NEU/LYM Ratio and Mortality Correlation | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  To investigate the prognostic role of the Neutrophil-to-Lymphocyte Ratio (NEU/LYM) (unit: ratio value) in predicting mortality among thoracic trauma patients. NEU/LYM values were obtained from complete blood count (CBC) results and recorded at 1st, 3rd, and 7th days
Glasgow Coma Scale (GCS) and Mortality Correlation | Measurements taken on day 1, day 3, and day 7 of hospitalization.
  Description: To evaluate the predictive value of the Glasgow Coma Scale (GCS) score on mortality and other clinical outcomes in thoracic trauma patients.
  Score Range: 3-15 (lower scores indicate worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: pınar karabacak, Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Determann RM, Royakkers AA, Haitsma JJ, Zhang H, Slutsky AS, Ranieri VM, Schultz MJ. Plasma levels of surfactant protein D and KL-6 for evaluation of lung injury in critically ill mechanically ventilated patients. BMC Pulm Med. 2010 Feb 16;10:6. doi: 10.1186/1471-2466-10-6. PMID 20158912
- [Background] Baker JE, Millar DA, Heh V, Goodman MD, Pritts TA, Janowak CF. Does chest wall Organ Injury Scale (OIS) or Abbreviated Injury Scale (AIS) predict outcomes? An analysis of 16,000 consecutive rib fractures. Surgery. 2020 Jul;168(1):198-204. doi: 10.1016/j.surg.2020.04.032. Epub 2020 May 13. PMID 32507628
- [Background] Lundin A, Akram SK, Berg L, Goransson KE, Enocson A. Thoracic injuries in trauma patients: epidemiology and its influence on mortality. Scand J Trauma Resusc Emerg Med. 2022 Dec 12;30(1):69. doi: 10.1186/s13049-022-01058-6. PMID 36503613